CLINICAL TRIAL: NCT02440659
Title: Empowering Patients on Choices for Renal Replacement Therapy (Aim 2)
Acronym: EPOCH-RRT
Status: Completed | Type: Observational
Sponsor: Arbor Research Collaborative for Health (Other)
Collaborators: University of Michigan (Other); Henry Ford Health System (Other); National Kidney Foundation, United States (Other); American Association of Kidney Patients (Other); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 1109201303132
Record Dates: First submitted 2015-04-09; First posted 2015-05-12 (Estimated); Results first posted 2016-10-04 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-04

CONDITIONS: Chronic Kidney Disease
Keywords: Chronic Kidney Disease; Hemodialysis; Peritoneal Dialysis
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Hemodialysis (HD): Patients who have chronic kidney disease (CKD) and are currently on hemodialysis.
- Peritoneal Dialysis (PD): Patients who have chronic kidney disease (CKD) and are currently on peritoneal dialysis.

SUMMARY:
Empowering Patients On Choices for Renal Replacement Therapy (EPOCH-RRT) study seeks to identify factors that matter the most to patients with kidney disease and study how they are impacted by different types of dialysis. The inclusion of patients, caregivers, and patient advocacy organizations as research partners will assure that the study addresses questions of greatest relevance to patients facing the need for dialysis.

Aim two is based on preliminary results of Aim one interviews, and in collaboration with the Patient Advisory Panel, the investigators developed a brief questionnaire to be administered to participants in the Dialysis Outcomes and Practice Patterns Study (DOPPS) and Peritoneal Dialysis Outcomes and Practice Patterns Study (PDOPPS). Two separate versions of the questionnaire were created to reflect unique aspects of in-center hemodialysis (HD) and peritoneal dialysis (PD).

ELIGIBILITY:
Inclusion Criteria:

* Individuals 18 years of age or older.
* Currently consented in the Dialysis Outcomes and Practice Patterns Study - (DOPPS) or the Peritoneal Outcomes and Practice Patterns Study (PDOPPS).

Exclusion Criteria:

* Individuals under 18 years of age.
* Individuals unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients currently consented in the Dialysis Outcomes and Practice Patterns Study (DOPPS) or the Peritoneal Outcomes and Practice Patterns Study (PDOPPS).
Sampling Method: Non-Probability Sample
Enrollment: 2946 (Actual)
Dates: Start 2015-02; Primary Completion 2015-08 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Tentori, MD, MS, Principal Investigator — Arbor Research Collaborative for Health
Locations (1):
- Arbor Research Collaborative for Health, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hemodialysis (HD) | Peritoneal Dialysis (PD)
Started | 1997 | 949
Completed | 1346 | 614
Not Completed | 651 | 335

BASELINE CHARACTERISTICS:
Population: Some baseline characteristics were missing for some participants. 10 participants were missing gender information and 12 participants were missing age information.
Groups:
- Total: Total of all reporting groups
Arm/Group | Hemodialysis (HD) | Peritoneal Dialysis (PD) | Total
Number analyzed (Participants) | 1346 | 614 | 1960
Age, Customized [Number; unit: participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 686 | 384 | 1070
  >=65 years | 649 | 229 | 878
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.04 (14.44) | 59.90 (14.92) | 62.06 (14.66)
Sex/Gender, Customized [Number; unit: participants]
  Female | 571 | 282 | 853
  Male | 766 | 331 | 1097
Region of Enrollment [Number; unit: participants]
  United States | 1346 | 614 | 1960

OUTCOME MEASURES:

1. Primary Outcome: Patient's Quality of Life
Description: % of patients very much or extremely affected by dialysis
Time Frame: Baseline
Measure: Number; unit: % of patients
Arm/Group | Hemodialysis (HD) | Peritoneal Dialysis (PD)
Number analyzed (Participants) | 1346 | 614
% of patients
  Relying on myself | 34 | 38
  Doing what I want in my free time | 35 | 27
  Spending time with people I care about | 34 | 21
  Doing activities that I am interested in | 28 | 21
  Traveling out of town | 45 | 42
  Maintaining a normal lifestyle | 27 | 24
  Managing my daily schedule | 21 | 17
  Keeping up with chores | 26 | 24
  Being energetic | 32 | 28
  Exercising | 22 | 20
  Maintaining my weight | 23 | 21
  Drinking as much water as I want | 46 | 24
  Eating what I like | 38 | 24
  Feeling healthy | 26 | 22
  Feeling attractive | 19 | 17
  Getting enough sleep | 26 | 22

ADVERSE EVENTS:
Description: Serious and Other [Not Including Serious] Adverse Events were not anticipated nor monitored/assessed.
Arm/Group | Hemodialysis (HD) | Peritoneal Dialysis (PD)
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No